CLINICAL TRIAL: NCT01556464
Title: Initiation of Auto-adjusting Continuous Positive Airway Pressure (CPAP) for Management of Newly Diagnosed Obstructive Sleep Apnea (OSA) in Hospitalized Patients: A Pilot Study
Brief Title: Initiation of Auto-adjusting CPAP for Newly Diagnosed OSA in Hospitalized Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with enrollment.
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Dennis Auckley, MD, Associate Professor of Medicine, Case Western Reserve University (CWRU), MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB11-00676
Record Dates: First submitted 2012-03-12; First posted 2012-03-16 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACPAP (Experimental): Patients in the intervention group will be introduced to the auto-adjusting CPAP (ACPAP) (ResMed S9) during the day and placed on it at night with a nocturnal oximetry and ACPAP download to assess its effectiveness and pressure requirements. The intervention is the application of the ACPAP. The patients will be discharged on ACPAP pressure determined by the ACPAP download (95th percentile pressure in absence of significant air leak) and will be scheduled for an outpatient repeat diagnostic PSG and, if indicated, a full night titration study.
  Interventions: Device: Auto-adjusting CPAP
- Control (No Intervention): The control group will receive nocturnal oxygen or no therapy while in the hospital and after discharge at the discretion of the attending physician. They will be scheduled for outpatient repeat diagnostic PSG and then, if indicated, a full night titration study.

INTERVENTIONS:
Device: Auto-adjusting CPAP — A CPAP device that auto-adjusts the pressure setting over the course of the night, depending on how the patient is breathing.
  Other Names: ResMed S9-Autoset CPAP
  Arms: ACPAP

SUMMARY:
This study will test the following hypotheses:

1. Treatment of newly diagnosed Obstructive Sleep Apnea (OSA) in acutely ill patients with auto-adjusting Continuous Positive Airway Pressure (CPAP) would result in fewer in-hospital complications, as compared to no treatment (primary outcome).
2. Treatment of newly identified OSA in acutely ill patients with auto-adjusting CPAP would result in shorter length of stay, lower re-admission rate, better blood pressure (BP) control, better long term compliance with OSA treatment, as compared to no treatment (secondary outcomes).

DETAILED DESCRIPTION:
This will be a pilot study performed as a randomized controlled prospective study of patients admitted to the general medical floors at MetroHealth Medical Center (MHMC). This study will be an add-on investigation to an original funded study: "Evaluation of Screening Tools for Obstructive Sleep Apnea (OSA) in Hospitalized Medical Patients: A Validation Study" (the STOMP study).

In the STOMP study, patients admitted Sunday through Thursday (day or night) to MHMC who meet inclusion/exclusion criteria and are willing to participate in the study will complete the STOMP study by undergoing an in-hospital PSG (within 48 hours of admission to the medical floor). Those who's PSG shows clinically significant OSA (an apnea-hypopnea index (AHI) > 5) will be approached for participation in this study. It is anticipated that at least 50 patients from the STOMP study will be eligible for randomization into this study. Participants will be randomized into an auto-adjusting Continuous Positive Airway Pressure (ACPAP) (ResMed S9) arm or a standard therapy arm (control - no specific therapy for OSA other than possibly supplemental nocturnal oxygen if deemed necessary by the clinicians caring for the patient). Those randomized to ACPAP will continue this therapy until they undergo a repeat diagnostic sleep study (PSG) and then, if indicated, a titration PSG as an outpatient. Those in the standard therapy arm will receive no specific treatment for their OSA until they undergo a a repeat diagnostic study and then, if indicated, a full night titration PSG as an outpatient. Once the titration PSG has taken place, subjects will be changed to fixed CPAP and followed for an additional 6-8 weeks to assess compliance with therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18-65 years old
* Admitted to the general medical floors on 6C, 9B, 10C, or 11C at MetroHealth Medical Center
* Expected stay of 48 hours
* Competent to sign informed consent
* Agreeable to participating in the study
* Underwent in-hospital PSG

Exclusion Criteria:

* Known OSA prior to admission
* Hypoventilation
* Patients with central sleep apnea
* Patients with a tracheostomy
* Clinically unstable patients with plans for transfer to a higher acuity of care
* Patients with planned surgical interventions or status post operation during the admission
* Patients transferred from intensive care
* Patients with respiratory failure requiring noninvasive ventilation
* Inability to comprehend or complete the questionnaires
* Inability to tolerate a sleep study (i.e. allergic to testing components, refusal to wear leads)
* Refusal to sign consent
* Non-English speaking patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
In-hospital complications | During hospitalization - anticipated average of 3 days
  Intubation, acute hypercapnia, need for supplemental oxygen, urgent respiratory support, Intensive Care Unit (ICU) transfer, arrhythmia, heart atack (MI), congestive heart failure (CHF), delerium, death

SECONDARY OUTCOMES:
CPAP compliance | 3 months
  CPAP compliance at 3 months after hospitalization
Length of stay | In-hospital time - expected average of 3 days
  Length of hospital stay
Readmission rate | 3 months after hospitalization
  90 day readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Auckley, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Goring K, Collop N. Sleep disordered breathing in hospitalized patients. J Clin Sleep Med. 2008 Apr 15;4(2):105-10. PMID 18468307
- [Background] Al-Jawder S, Bahammam A. Utility of daytime polysomnography for in-patients with suspected sleep-disordered breathing. Neurol Neurochir Pol. 2009 Mar-Apr;43(2):140-7. PMID 19484691
- [Background] Padeletti M, Green P, Mooney AM, Basner RC, Mancini DM. Sleep disordered breathing in patients with acutely decompensated heart failure. Sleep Med. 2009 Mar;10(3):353-60. doi: 10.1016/j.sleep.2008.03.010. Epub 2008 Jul 9. PMID 18614398
- [Background] Spurr KF, Graven MA, Gilbert RW. Prevalence of unspecified sleep apnea and the use of continuous positive airway pressure in hospitalized patients, 2004 National Hospital Discharge Survey. Sleep Breath. 2008 Aug;12(3):229-34. doi: 10.1007/s11325-007-0166-2. Epub 2008 Jan 31. PMID 18236092
- [Background] Khayat RN, Abraham WT, Patt B, Pu M, Jarjoura D. In-hospital treatment of obstructive sleep apnea during decompensation of heart failure. Chest. 2009 Oct;136(4):991-997. doi: 10.1378/chest.09-0597. Epub 2009 Jun 30. PMID 19567491
- [Background] Nader NZ, Steinel JA, Auckley DH. Newly identified obstructive sleep apnea in hospitalized patients: analysis of an evaluation and treatment strategy. J Clin Sleep Med. 2006 Oct 15;2(4):431-7. PMID 17557473